CLINICAL TRIAL: NCT06333496
Title: Effect of a Glucagon Like Peptide 1 (GLP1) Booster on Blood Glucose, HbA1c, Insulin, and GLP1 Levels, Body Weight and Body Fat in Overweight Adult Men and Women
Brief Title: Effect of a Glucagon Like Peptide 1 (GLP1) Booster in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alpine Biotech LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB20240102H
Record Dates: First submitted 2024-03-11; First posted 2024-03-27 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-06

CONDITIONS: Blood Sugar; High; Overweight and Obesity; Fat Burn; Obesity; Heart Health Markers
MeSH Terms: conditions — Hyperglycemia; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GLP-1 Booster (Experimental): GLP-1 Booster (GB) is a composition designed to increase the endogenous production of GLP-1, improve the activity of GLP-1, enhance the body's response to GLP-1, and thus eventually help people reduce glucose, suppress food intake and lose body fat. GB contains Green tea (Camellia sinensis) leaf extract, Gardeniae (Gardenia jasminoides Ellis) fructus extract, Turmeric (Curcuma longa) root extract, Black pepper (Piper nigrum) extract,Fenugreek (Trigonella foenum-graecum) seed extract, Ginseng (Panax ginseng) root extract, and White kidney bean (Phaseolus vulgaris) extract. Each of these ingredients has been commonly consumed by humans as food sources or supplements and thus has an undebatable safety profile.
  Interventions: Dietary Supplement: GLP-1 Booster (GB)

INTERVENTIONS:
Dietary Supplement: GLP-1 Booster (GB) — GLP-1 Booster (GB) is a composition designed to increase the endogenous production of GLP-1, improve the activity of GLP-1, enhance the body's response to GLP-1, and thus eventually help people reduce glucose, suppress food intake and lose body fat. GB contains Green tea (Camellia sinensis) leaf extract, Gardeniae (Gardenia jasminoides Ellis) fructus extract, Turmeric (Curcuma longa) root extract, Black pepper (Piper nigrum) extract,Fenugreek (Trigonella foenum-graecum) seed extract, Ginseng (Panax ginseng) root extract, and White kidney bean (Phaseolus vulgaris) extract. Each of these ingredients has been commonly consumed by humans as food sources or supplements and thus has an undebatable safety profile.

SUMMARY:
BACKGROUND GLP1 booster (GB) was designed to stimulate the endogenous production of GLP1, which in turn releases insulin, controls blood glucose level, suppresses appetite and thus helps people lose weight.

PURPOSE The purpose of this study is to assess several clinical endpoints and questionnaires in healthy volunteers taking the new GB formula.

SCOPE The scope of this protocol covers the non-clinical portion as well as the assessment of several clinical endpoints and questionnaires. In brief, the non-clinical design will be an open-label study involving volunteers taking GB everyday for 12 weeks. Data analysis will involve measuring the clinical endpoints across the group at different timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must be over the age of 18.
* Volunteers cannot be smokers.
* Volunteers cannot be currently taking a dietary supplement or prescription for weight loss.
* Exercising volunteers must maintain their regimen consistently throughout the course of the 12-week study.
* Caffeine drinking volunteers must maintain their caffeine intake consistently throughout the course of the 12-week study.
* Volunteers need to be overweight but not obese, as defined by having a BMI between 25.0 and 29.9

Exclusion Criteria:

* Female volunteers who are pregnant or planning to become pregnant within the next three months.
* Volunteers who are taking any stimulant medications (e.g. Adderall, Adzenys, Dexedrine, Ritalin, Methylphenidate, etc).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
blood glucose level | 12 week
blood HbA1c level | 12 week
blood insulin level | 12 week
blood GLP1 level | 12 week
blood cholesterol level | 12 week
body weight | 12 week
body fat mass | 12 week
body lean mass | 12 week
body mass index | 12 week
body fat index | 12 week
waist hip ratio | 12 week

SECONDARY OUTCOMES:
Satiety score | 12 week
Resting metabolic rate | 12 week
Blood pressure | 12 week
  both systolic and diastolic pressures
Heart rate | 12 week

CONTACTS AND LOCATIONS:
Overall Officials: Lawry Han, PhD, Principal Investigator — Alpine Biotech LLC
Locations (1):
- Alpine Bio, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No